CLINICAL TRIAL: NCT00105989
Title: Duloxetine Versus Placebo in the Prevention of Recurrence of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8606; F1J-MC-HMDI
Record Dates: First submitted 2005-03-18; First posted 2005-03-21 (Estimated); Results first posted 2009-07-17 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Experimental): duloxetine 60-120 mg every day (QD), by mouth (PO) for 34 weeks followed by duloxetine 60-120 mg QD, PO for up to 54 weeks
  Interventions: Drug: Duloxetine
- B (Placebo Comparator): duloxetine 60-120 mg every day (QD), by mouth (PO) for 34 weeks followed by placebo QD, PO for up to 54 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Duloxetine
  Other Names: LY248686; Cymbalta
  Arms: A
Drug: placebo
  Arms: B

SUMMARY:
The purpose of this study is to assess the efficacy and safety of duloxetine compared with placebo in the prevention of depressive recurrences among patients with recurrent major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years old.
* Patient must be diagnosed with depression and have had previous episodes of depression.
* Patient must sign informed consent.

Exclusion Criteria:

* Female and pregnant or breastfeeding.
* History of bipolar disorder, schizophrenia, or other psychotic disorders.
* Suffer from a serious medical illness (other than depression) or abnormal laboratory result that would require a change in medication, intervention, or hospitalization.
* Have been treated with a medication called monoamine oxidase inhibitor (MAOI) within 14 days of the start of the study, or potential need to use a MAOI within 5 days of finishing the study.
* Have taken an antidepressant called fluoxetine within 30 days of the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2005-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (34):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherman Oaks, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaithersburg, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
- France (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Angoulême
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Douai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fains
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Rochelle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roubaix
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ellwangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hildesheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Würzburg
- Italy (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ferrara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Village Nikolskoe
- Sweden (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halmstad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sundsvall

REFERENCES:
- [Derived] Perahia DG, Maina G, Thase ME, Spann ME, Wang F, Walker DJ, Detke MJ. Duloxetine in the prevention of depressive recurrences: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2009 May;70(5):706-16. doi: 10.4088/jcp.08m04756. PMID 19552867
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Acute - Open Label (Week 0-10) participants were reported in the Baseline Characteristics section of this results record.
Groups:
- Duloxetine: duloxetine 60-120 mg every day (QD), by mouth (PO) for 34 weeks followed by duloxetine 60-120 mg QD, PO for up to 54 weeks.
- Placebo: duloxetine 60-120 mg every day (QD), by mouth (PO) for 34 weeks followed by placebo QD, PO for up to 54 weeks.
Period: Acute - Open Label: Week 0-10
Arm/Group | Duloxetine | Placebo
Started | 514 | 0
Completed | 413 | 0
Not Completed | 101 | 0
Not completed — Adverse Event | 33 | 0
Not completed — Withdrawal by Subject | 24 | 0
Not completed — Lack of Efficacy | 17 | 0
Not completed — Protocol Response Criteria Not Met | 14 | 0
Not completed — Protocol Violation | 8 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Physician Decision | 0 | 0
Not completed — Death | 1 | 0
Not completed — Recurrence Criteria Met | 0 | 0
Not completed — Unspecified - no reason reported | 0 | 0
Period: Continuation - Open Label:Week 10-34
Arm/Group | Duloxetine | Placebo
Started | 413 | 0
Completed | 288 | 0
Not Completed | 125 | 0
Not completed — Adverse Event | 25 | 0
Not completed — Withdrawal by Subject | 50 | 0
Not completed — Lack of Efficacy | 15 | 0
Not completed — Protocol Response Criteria Not Met | 16 | 0
Not completed — Protocol Violation | 5 | 0
Not completed — Lost to Follow-up | 9 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Death | 0 | 0
Not completed — Recurrence Criteria Met | 2 | 0
Not completed — Unspecified - no reason reported | 0 | 0
Period: Maintenance - Double-Blind:Week 34-86
Arm/Group | Duloxetine | Placebo
Started | 146 | 142
Completed | 96 | 73
Not Completed | 50 | 69
Not completed — Adverse Event | 6 | 3
Not completed — Withdrawal by Subject | 17 | 18
Not completed — Lack of Efficacy | 0 | 0
Not completed — Protocol Response Criteria Not Met | 0 | 0
Not completed — Protocol Violation | 5 | 4
Not completed — Lost to Follow-up | 4 | 0
Not completed — Physician Decision | 4 | 1
Not completed — Death | 0 | 0
Not completed — Recurrence Criteria Met | 14 | 43
Not completed — Unspecified - no reason reported | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Duloxetine: duloxetine 60-120 mg QD
Arm/Group | Duloxetine
Number analyzed (Participants) | 514
Age Continuous [Mean (Standard Deviation); unit: years] | 47.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 359
  Male | 155
Region of Enrollment [Number; unit: participants]
  United States | 61
  France | 65
  Russian Federation | 99
  Germany | 161
  Italy | 73
  Sweden | 55
Race/Ethnicity [Number; unit: participants]
  Caucasian | 504
  Hispanic | 5
  African | 3
  South Asian | 1
  East Asian | 1
17-item Hamilton Depression Rating Scale (HAMD-17) Total Score [Mean (Standard Deviation); unit: units on a scale] — The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (absent, mild, moderate, severe, very severe) or a 3-point scale (absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
  units on a scale | 23.07 (3.57)
Age at First Episode [Mean (Standard Deviation); unit: years] | 33.16 (13.38)
Clinical Global Impressions - Severity (CGI-S) Total Score [Mean (Standard Deviation); unit: units on a scale] — Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  units on a scale | 4.49 (0.6)
Duration of Current Episode [Mean (Standard Deviation); unit: months] | 4.02 (4.65)
Duration of Last Episode [Mean (Standard Deviation); unit: months] | 6.14 (5.29)
Height [Mean (Standard Deviation); unit: centimeters] | 167.6 (9.23)
Number of Previous Episodes [Mean (Standard Deviation); unit: previous episodes] | 4.22 (3.48)
Time Interval Between Episodes [Mean (Standard Deviation); unit: months] | 8.38 (6.78)
Weight [Mean (Standard Deviation); unit: kilograms] | 74.7 (16.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Depressive Recurrence After Time (t) in Days
Description: Recurrence: Clinical Global Impression-Severity (CGI-S) score >=4 and met Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for major depressive disorder (MDD); had 3 consecutive visits where re-emergence criteria met; had total of 10 visits where re-emergence criteria was satisfied; discontinued due to lack of efficacy.
Time Frame: Every Visit from Week 34 up to Week 86 (Maintenance Phase)
Population: All randomized patients. Intent to Treat analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 146 | 142
percentage of participants
  t=7 days (N=145, N=139) | 0.68 | 2.11
  t=14 days (N=143, N=138) | 1.37 | 2.11
  t=21 days (N=141, N=137) | 1.37 | 2.82
  t=28 days (N=140, N=135) | 2.07 | 3.54
  t=56 days (N=136, N=120) | 4.19 | 12.97
  t=84 days (N=131, N=106) | 6.33 | 21.15
  t=112 days (N=122, N=96) | 8.58 | 25.79
  t=140 days (N=119, N=89) | 9.34 | 28.98
  t=168 days (N=115, N=86) | 10.89 | 28.98
  t=196 days (N=111, N=86) | 11.69 | 28.98
  t=224 days (N=108, N=85) | 12.50 | 29.80
  t=252 days (N=105, N=82) | 13.32 | 32.28
  t=280 days (N=99, N=77) | 13.32 | 34.00
  t=308 days (N=96, N=75) | 13.32 | 34.86
  t=336 days (N=95, N=74) | 14.23 | 34.86
  t=364 days (N=93, N=73) | 16.03 | 35.74
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; A total of 257 randomized patients (randomly assigned with equal probability to the two treatment groups) were needed to have 90% power to detect 40% versus 20% recurrence rates over 52 weeks, using a log rank test at a two-sided significance level of .05; Test type: Superiority or Other; p < 0.001, Log Rank — No adjustments were made for multiple comparisons. The primary efficacy analysis compared the time to recurrence during the maintenance phase between all duloxetine and placebo patients using the log-rank test, stratified by country at α=.05; The log rank method provides a single p-value comparing time to depressive recurrence for placebo and duloxetine

2. Secondary Outcome: Recurrence Count
Description: Number of participants who experienced a depressive recurrence at any time during the double-blind maintenance therapy phase.
Time Frame: Every Visit from Week 35 up to Week 86 (Maintenance Phase)
Population: Number of randomized patients with at least one non-missing postbaseline assessment during the double-blind maintenance therapy phase. Intent to Treat analysis.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 146 | 142
participants | 21 | 47
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Frequencies are analyzed using Cochran-Mantel-Haenszel controlling for investigator

3. Secondary Outcome: Percentage of Participants With Greater Than or Equal to 50% Worsening After Time (t) in Days
Description: Worsening occurs if patient had a >=50% increase from baseline on the 17-Item Hamilton Depression Rating Scale (HAMD-17) total score and a Clinical Global Impression-Severity (CGI-S) score >=3 at any time during the double-blind maintenance therapy phase.
Time Frame: Every Visit from Week 34 up to Week 86 (Maintenance Phase)
Population: Number of randomized patients with at least one non-missing post-baseline assessment during the double blind maintenance therapy phase. Intent to Treat analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 146 | 142
percentage of participants
  t=7 days (N=142, N=140) | 2.07 | 1.41
  t=14 days (N=140, N=138) | 3.45 | 1.41
  t=21 days (N=136, N=130) | 5.53 | 7.12
  t=28 days (N=132, N=125) | 7.63 | 9.30
  t=56 days (N=124, N=105) | 11.89 | 22.57
  t=84 days (N=114, N=88) | 16.99 | 31.86
  t=112 days (N=105, N=81) | 21.48 | 35.07
  t=140 days (N=100, N=72) | 23.02 | 40.82
  t=168 days (N=95, N=70) | 24.61 | 42.47
  t=196 days (N=93, N=67) | 26.19 | 44.14
  t=224 days (N=90, N=65) | 28.57 | 45.80
  t=252 days (N=84, N=60) | 31.04 | 45.80
  t=280 days (N=81, N=60) | 31.88 | 45.80
  t=308 days (N=78, N=59) | 31.88 | 46.71
  t=336 days (N=77, N=56) | 31.88 | 49.42
  t=364 days (N=75, N=51) | 33.65 | 51.33
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, Log Rank; The log rank method provides a single p-value comparing time to depressive recurrence for placebo and duloxetine

4. Secondary Outcome: Loss of Response at Any Time
Description: Loss of response was defined as a HAMD-17 total score >9 and a CGI-Severity score >2 at any one time during the double-blind maintenance phase of the study regardless of whether or not they subsequently regained response or not.
Time Frame: Every Visit from Week 35 up to Week 86 (Maintenance Phase)
Population: Number of randomized patients with at least one non-missing post-baseline assessment during the double-blind maintenance therapy phase. Intent to Treat analysis.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 146 | 142
participants | 44 | 66
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel; Frequencies were analyzed using Cochran-Mantel-Haenszel controlling for investigator

5. Secondary Outcome: Change From Baseline to Endpoint in 17-Item Hamilton Depression Rating Scale (HAMD-17) Total Score - Acute and Continuation Phases
Description: The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: Number of enrolled patients in the Acute Phase with a baseline and at least one non-missing post-baseline measurement. Number of patients who entered Continuation phase with baseline and have at least 1 post-baseline measurement. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Duloxetine - Acute Phase: duloxetine 60-120 mg every day (QD) from Week 0 (baseline) to Week 10 (Endpoint)
- Duloxetine - Continuation Phase: duloxetine 60-120 mg every day (QD) from Week 10 (baseline) to Week 34 (Endpoint)
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 503 | 412
units on a scale
  Baseline | 23.07 (3.55) | 6.64 (2.06)
  Change from Baseline to Endpoint | -14.37 (6.03) | -0.61 (5.09)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.016, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

6. Secondary Outcome: Change From Baseline to Endpoint in 17-Item Hamilton Depression Rating Scale (HAMD-17) Total Score - Maintenance Phase
Description: The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (absent, mild, moderate, severe, very severe) or a 3-point scale (absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline measurement. Intent to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 145 | 142
units on a scale | 1.40 (0.53) | 4.36 (0.57)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

7. Secondary Outcome: Change From Baseline to Endpoint in Clinical Global Impressions (CGI) Severity Scale - Acute and Continuation Phases
Description: Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 503 | 412
units on a scale
  Baseline | 4.49 (0.60) | 1.83 (0.39)
  Change from Baseline to Endpoint | -2.30 (1.08) | -0.07 (0.93)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.153, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

8. Secondary Outcome: Change From Baseline to Endpoint in Clinical Global Impressions (CGI) Severity Scale - Maintenance Phase
Description: Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients.
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline assessment. Intent to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 145 | 142
units on a scale | 0.24 (0.10) | 0.84 (0.10)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

9. Secondary Outcome: Mean Values at Endpoint in Patient's Global Impressions of Improvement (PGI-I) - Acute and Continuation Phases
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: Week 10 (Acute) and Week 34 (Continuation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 488 | 412
units on a scale | 2.12 (0.86) | 1.76 (0.91)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; t-test assesses if within treatment mean value at endpoint is significant from 4
Statistical Analysis 2: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; t-test assesses if within treatment mean value at endpoint is significant from 4

10. Secondary Outcome: Mean Values at Endpoint in Patient's Global Impressions of Improvement (PGI-I) - Maintenance Phase
Description: as for outcome 9
Time Frame: Week 86 (Maintenance Phase)
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 145 | 142
units on a scale | 1.72 (0.11) | 2.34 (0.11)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

11. Secondary Outcome: Change From Baseline to Endpoint in Hamilton Depression Rating Scale Subscales, Including the Core, Maier, Anxiety/Somatization, Retardation/Somatization, and Sleep Subscales, and the Depressed Mood Item - Acute and Continuation Phases
Description: Core and Maier subscales assess symptoms of depression (scores:0-20=Core; 0-24=Maier). Higher numbers indicate more severe symptoms. Anxiety/Somatization subscale assesses severity of anxiety (0-18). Retardation subscale assesses dysfunction in mood and work (0-14). Sleep subscale assesses insomnia (0-6). Depressed Mood Item (0-4).
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 503 | 412
units on a scale
  Anxiety Baseline | 7.71 (1.99) | 2.51 (1.40)
  Anxiety Change from Baseline to Endpoint | -4.52 (2.63) | -0.11 (2.24)
  Core Baseline | 8.81 (1.78) | 2.00 (1.35)
  Core Change from Baseline to Endpoint | -5.97 (2.69) | -0.29 (2.47)
  Maier Baseline | 11.44 (1.95) | 2.91 (1.60)
  Maier Change from Baseline to Endpoint | -7.46 (3.29) | -0.29 (2.97)
  Retardation Baseline | 7.76 (1.53) | 2.43 (1.37)
  Retardation Change from Baseline to Endpoint | -4.61 (2.37) | -0.48 (2.22)
  Sleep Baseline | 3.80 (1.59) | 1.11 (1.11)
  Sleep Change from Baseline to Endpoint | -2.37 (1.92) | -0.07 (1.38)
  Depressed Mood Baseline | 2.78 (0.58) | 0.64 (0.57)
  Depressed Mood Change from Baseline to Endpoint | -1.86 (0.98) | -0.05 (0.95)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-values for Change from Baseline to Endpoint for all Subscales during Acute phase were <0.001; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.334, t-test, 2 sided — P-value for Anxiety Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 3: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.019, t-test, 2 sided — P-value for Core Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 4: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.046, t-test, 2 sided — P-value for Maier Change from Baseline to Endpoint; t-test assessses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 5: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Retardation Change from Baseline to Endpoint; t-test assessses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 6: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.319, t-test, 2 sided — P-value for Sleep Change from Baseline to Endpoint; t-test assessses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 7: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.275, t-test, 2 sided — P-value for Depressed Mood Change from Baseline to Endpoint; t-test assessses if within treatment mean changes from baseline to endpoint are significantly different from zero

12. Secondary Outcome: Change From Baseline to Endpoint in Hamilton Depression Rating Scale Subscales, Including the Core, Maier, Anxiety/Somatization, Retardation/Somatization, and Sleep Subscales, and the Depressed Mood Item - Maintenance Phase
Description: as for outcome 11
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 145 | 142
units on a scale
  Change from Baseline to Endpoint in Anxiety | 0.46 (0.20) | 1.54 (0.22)
  Change from Baseline to Endpoint in Core | 0.75 (0.22) | 1.74 (0.24)
  Change from Baseline to Endpoint in Maier | 0.91 (0.29) | 2.25 (0.31)
  Change from Baseline to Endpoint in Retardation | 0.59 (0.20) | 1.49 (0.22)
  Change from Baseline to Endpoint in Sleep | 0.13 (0.12) | 0.71 (0.13)
  Change from Baseline to Endpoint in Depressed Mood | 0.27 (0.09) | 0.67 (0.10)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Pairwise comparison of Least Squares Means for Anxiety Subscale Change from Baseline to Endpoint
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 2 sided — P-value for Pairwise comparison of Least Squares Means for Core Subscale Change from Baseline to Endpoint
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 2 sided — P-value for Pairwise comparison of Least Squares Means for Maier Subscale Change from Baseline to Endpoint
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, t-test, 2 sided — P-value for Pairwise comparison of Least Squares Means for Retardation Subscale Change from Baseline to Endpoint
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — P-value for Pairwise comparison of Least Squares Means for Sleep Subscale Change from Baseline to Endpoint
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, t-test, 2 sided — P-value for Pairwise comparison of Least Squares Means for Depressed Mood Subscale Change from Baseline to Endpoint

13. Secondary Outcome: Change From Baseline to Endpoint in Visual Analog Scales (VAS) for Pain - Acute and Continuation Phase
Description: VAS for pain consists of 6 questions that assess overall pain, headache, back pain, shoulder pain, pain interference with daily activities, and pain while awake. Participant rates pain on a 100 millimeter (mm) line between two anchors (0 = no pain and 100 = very severe pain).
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 450 | 410
units on a scale
  Overall Pain Baseline (N=450, N=410) | 34.36 (26.16) | 17.29 (20.20)
  Overall Pain Change from Baseline to Endpoint | -16.34 (26.95) | 1.16 (21.33)
  Headache Baseline (N=450, N=410) | 29.74 (28.08) | 14.80 (20.53)
  Headache Change from Baseline to Endpoint | -14.83 (28.04) | 0.04 (21.88)
  Back Pain Baseline (N=450, N=410) | 28.79 (27.80) | 15.61 (22.63)
  Back Pain Change from Baseline to Endpoint | -13.64 (25.66) | -0.00 (20.95)
  Shoulder Pain Baseline (N=446, N=410) | 24.06 (27.23) | 13.49 (21.95)
  Shoulder Pain Change from Baseline to Endpoint | -10.47 (24.25) | -0.39 (20.84)
  Interference-DailyActivities Baseline(N=445,N=410) | 33.28 (28.31) | 15.59 (21.62)
  Intereference Change from Baseline to Endpoint | -16.79 (29.77) | 1.00 (21.43)
  Pain While Awake Baseline (N=446, N=410) | 38.18 (29.29) | 19.22 (25.63)
  Pain While Awake Change from Baseline to Endpoint | -17.66 (31.22) | 0.06 (25.61)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for all Change from Baseline to Endpoint measures in the Acute Phase were <0.001; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.273, t-test, 2 sided — P-value for Overall Pain Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 3: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.968, t-test, 2 sided — P-value for Headache Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 4: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.998, t-test, 2 sided — P-value for Back Pain Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 5: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.703, t-test, 2 sided — P-value for Shoulder Pain Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 6: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.346, t-test, 2 sided — P-value for Interference with Daily Activities Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 7: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.963, t-test, 2 sided — P-value for Pain While Awake Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

14. Secondary Outcome: Change From Baseline to Endpoint in Visual Analog Scales (VAS) for Pain - Maintenance Phase
Description: as for outcome 13
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 146 | 142
units on a scale
  Change from Baseline to Endpoint in Overall Pain | 3.92 (1.78) | 4.57 (1.86)
  Change from Baseline to Endpoint in Headache | 4.77 (1.72) | 2.80 (1.80)
  Change from Baseline to Endpoint in Back Pain | 1.77 (1.65) | 3.40 (1.72)
  Change from Baseline to Endpoint in Shoulder Pain | 0.51 (1.55) | 3.02 (1.62)
  Change: Interference with Daily Activities | 3.16 (1.74) | 2.81 (1.82)
  Change from Baseline in Pain While Awake | 3.64 (2.10) | 4.69 (2.19)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.792, t-test, 2 sided — P-value for pairwise comparison of Least Squares Means for Overall Pain Change from Baseline to Endpoint
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.407, t-test, 2 sided — P-value for pairwise comparison of Least Squares Means for Headache Change from Baseline to Endpoint
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.475, t-test, 2 sided — P-value for pairwise comparison of Least Squares Means for Back Pain Change from Baseline to Endpoint
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.241, t-test, 2 sided — P-value for pairwise comparison of Least Squares Means for Shoulder Pain Change from Baseline to Endpoint
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.885, t-test, 2 sided — P-value for pairwise comparison of Least Squares Means for Interference with Daily Activities Change from Baseline to Endpoint
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.717, t-test, 2 sided — P-value for pairwise comparison of Least Squares Means for Pain While Awake Change from Baseline to Endpoint

15. Secondary Outcome: Change From Baseline to Endpoint in Symptom Questionnaire-Somatic Subscale (SQ-SS) - Acute and Continuation Phases
Description: The Somatic subscale consists of 23 items to be completed by the patient that focus on somatic symptoms. Question answers are either yes/no or true/false. Negative response is scored at 1; positive response is scored as 0. Total Somatic subscale scores range from 0-23, where higher scores indicate greater symptom severity.
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 448 | 376
units on a scale
  Baseline | 12.64 (5.09) | 6.88 (5.13)
  Change from Baseline to Endpoint | -5.37 (5.42) | -0.35 (4.80)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.157, t-test, 2 sided — P-value for Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

16. Secondary Outcome: Change From Baseline to Endpoint in Symptom Questionnaire-Somatic Subscale (SQ-SS) - Maintenance Phase
Description: as for outcome 15
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: Number of randomized patients with non-missing baseline and at least one non-missing post-baseline measurement. Intent to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 145 | 140
units on a scale | 0.79 (0.39) | 0.81 (0.40)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.979, t-test, 2 sided

17. Secondary Outcome: Change From Baseline to Endpoint in Sheehan Disability Scale (SDS) - Acute and Continuation Phases
Description: The SDS is completed by the patient and is used to assess the effect of the patient's symptoms on their work/social/family life. Total (Global) scores range from 0 to 30 with higher values indicating greater disruption in the patient's work/social/family life. Individual Item scores range from 0 to 10.
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 452 | 378
units on a scale
  Global Score Baseline (N=449,N=378) | 19.30 (6.58) | 10.72 (7.21)
  Global Score Change from Baseline to Endpoint | -7.88 (8.06) | -2.01 (7.67)
  Work/School Item Baseline (N=452,N=378) | 6.52 (2.52) | 3.64 (2.64)
  Work/School Item Change from Baseline to Endpoint | -2.61 (2.87) | -0.71 (2.86)
  Social Life Item Baseline (N=452,N=378) | 6.45 (2.42) | 3.50 (2.53)
  Social Life Item Change from Baseline to Endpoint | -2.69 (2.90) | -0.64 (2.79)
  Family Life Item Baseline (N=452,N=378) | 6.35 (2.44) | 3.54 (2.57)
  Family Life Item Change from Baseline to Endpoint | -2.59 (3.07) | -0.63 (2.72)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Change from Baseline to Endpoint in all SDS items in Acute Phase were <0.001; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Change from Baseline to Endpoint in all SDS items in the Continuation Phase were <0.001; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

18. Secondary Outcome: Change From Baseline to Endpoint in Sheehan Disability Scale (SDS) - Maintenance Phase
Description: as for outcome 17
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 128 | 117
units on a scale
  Change from Baseline to Endpoint in Global Score | -0.05 (0.71) | 2.06 (0.77)
  Change from Baseline to Endpoint in Work/School | 0.03 (0.26) | 0.83 (0.28)
  Change from Baseline to Endpoint in Social Life | 0.02 (0.25) | 0.56 (0.27)
  Change from Baseline to Endpoint in Family Life | -0.10 (0.25) | 0.67 (0.27)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.029, t-test, 2 sided — P-value for pairwise comparison of Least Squares Means for Change from Baseline to Endpoint in Global Score
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.022, t-test, 2 sided — P-value for pairwise comparison of Least Squares Means for Change from Baseline to Endpoint in Work/School
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.110, t-test, 2 sided — P-value for pairwise comparison of Least Squares Means for Change from Baseline to Endpoint in Social Life
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.021, t-test, 2 sided — P-value for pairwise comparison of Least Squares Means for Change from Baseline to Endpoint in Family Life/Home Responsibilities

19. Secondary Outcome: Change From Baseline to Endpoint in 36-item Short-Form Health Survey (SF-36) - Acute and Continuation Phase
Description: Assesses general quality of life. 36 questions covering 8 health domains. Each subscale is scored by summing the individual items and transforming scores into a 0-100 scale, with higher scores indicating better health status or functioning.
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 460 | 377
units on a scale
  Physical Component Summary Baseline (N=455,N=377) | 43.55 (9.46) | 48.05 (8.65)
  Physical Component Summary Change to Endpoint | 3.86 (8.66) | 0.03 (7.63)
  Mental Component Summary Baseline (N=455,N=377) | 23.93 (8.76) | 39.83 (10.68)
  Mental Component Summary Change to Endpoint | 14.67 (11.77) | 3.98 (12.63)
  Physical Functioning Baseline (N=457,N=377) | 23.59 (4.75) | 26.28 (4.05)
  Physical Functioning Change to Endpoint | 2.39 (4.40) | 0.28 (3.42)
  Bodily Pain Baseline (N=460,N=377) | 6.83 (2.45) | 8.61 (2.35)
  Bodily Pain Change from Baseline to Endpoint | 1.61 (2.50) | 0.07 (2.39)
  Role Limitations:Physical Baseline (N=457,N=377) | 5.24 (1.47) | 6.48 (1.54)
  Role Limitations:Physical Change to Endpoint | 1.06 (1.78) | 0.20 (1.74)
  Role Limitations:Emotional Baseline (N=456,N=377) | 3.42 (0.80) | 4.65 (1.25)
  Role Limitations:Emotional Change to Endpoint | 1.11 (1.31) | 0.34 (1.49)
  General Health Perceptions Baseline(N=456,N=377) | 13.66 (3.62) | 17.03 (3.80)
  General Health Perceptions Change to Endpoint | 2.93 (3.74) | 0.58 (3.52)
  Mental Health Baseline (N=456,N=377) | 12.62 (4.13) | 19.60 (4.39)
  Mental Health Change from Baseline to Endpoint | 6.45 (5.31) | 1.30 (5.34)
  Social Function Baseline (N=460,N=377) | 4.77 (1.74) | 7.05 (1.80)
  Social Function Change from Baseline to Endpoint | 2.12 (2.04) | 0.65 (2.19)
  Vitality Baseline (N=457,N=377) | 8.85 (3.26) | 13.84 (3.79)
  Vitality Change from Baseline to Endpoint | 4.51 (4.22) | 0.84 (4.40)
  Rate Current Health Baseline (N=460,N=377) | 3.88 (0.85) | 3.03 (0.83)
  Rate Current Health Change to Endpoint | -0.72 (0.95) | -0.01 (0.88)
  Health Compared to Year Ago Baseline (N=460,N=377) | 3.67 (0.99) | 2.37 (1.05)
  Health Compared to Year Ago Change to Endpoint | -1.18 (1.28) | -0.34 (1.13)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-values for Change from Baseline to Endpoint in all SF-36 subscales in the Acute Phase were <0.001; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.947, t-test, 2 sided — P-value for Physical Component Summary Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 3: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Mental Component Summary Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 4: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.118, t-test, 2 sided — P-value for Physical Functioning Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 5: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.550, t-test, 2 sided — P-value for Bodily Pain Change from Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 6: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.029, t-test, 2 sided — P-value for Role Limitations Due to Physical Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 7: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Role Limitations Due to Emotional Problems Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 8: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.002, t-test, 2 sided — P-value for General Health Perceptions Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 9: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Mental Health Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 10: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Social Function Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 11: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Vitality Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 12: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.815, t-test, 2 sided — P-value for Rate Current Health Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 13: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Health Compared to a Year Ago Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

20. Secondary Outcome: Change From Baseline to Endpoint in 36-item Short-Form Health Survey (SF-36) - Maintenance Phase
Description: as for outcome 19
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 129 | 118
units on a scale
  Change from Baseline-Physical Component Summary | -0.45 (0.70) | 0.33 (0.76)
  Change from Baseline-Mental Component Summary | -1.11 (1.11) | -5.74 (1.20)
  Change from Baseline-Physical Functioning | 0.06 (0.28) | -0.07 (0.31)
  Change from Baseline-Bodily Pain | -0.42 (0.22) | -0.19 (0.24)
  Change from Baseline-Role Limitations: Physical | 0.01 (0.14) | -0.41 (0.15)
  Change from Baseline-Role Limitations: Emotional | -0.03 (0.11) | -0.46 (0.11)
  Change from Baseline-General Health Perceptions | -0.23 (0.33) | -0.61 (0.36)
  Change from Baseline-Mental Health | -0.44 (0.49) | -2.60 (0.53)
  Change from Baseline-Social Function | -0.14 (0.18) | -0.50 (0.20)
  Change from Baseline-Vitality | -0.77 (0.38) | -1.38 (0.41)
  Change from Baseline-Rate Current Health | 0.03 (0.08) | 0.08 (0.08)
  Change from Baseline-Health Compared to Year Ago | 0.19 (0.09) | 0.34 (0.10)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.415, t-test, 2 sided — P-value is pairwise comparison of Least Squares Means for Change from Baseline-Physical Component Summary
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 2 sided — P-value is pairwise comparison of Least Squares Means for Change from Baseline-Mental Component Summary
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.731, t-test, 2 sided — P-value is pairwise comparison of Least Squares Means for Change from Baseline-Physical Functioning
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.438, t-test, 2 sided — P-value is pairwise comparison of Least Squares Means for Change from Baseline-Bodily Pain
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.029, t-test, 2 sided — P-value is pairwise comparison of Least Squares Means for Change from Baseline-Role Limitations Due to Physical
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, t-test, 2 sided — P-value is pairwise comparison of Least Squares Means for Change from Baseline-Role Limitations Due to Emotional problems
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.391, t-test, 2 sided — P-value is pairwise comparison of Least Squares Means for Change from Baseline-General Health Perceptions
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — P-value is pairwise comparison of Least Squares Means for Change from Baseline-Mental Health
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.142, t-test, 2 sided — P-value is pairwise comparison of Least Squares Means for Change from Baseline-Social Functioning
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.240, t-test, 2 sided — P-value is pairwise comparison of Least Squares Means for Change from Baseline-Vitality
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.615, t-test, 2 sided — P-value is pairwise comparison of Least Squares Means for Change from Baseline-Rate General Health
Statistical Analysis 12: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.218, t-test, 2 sided — P-value is pairwise comparison of Least Squares Means for Change from Baseline-Health Compared to a Year Ago

21. Secondary Outcome: Resource Utilization and Hospitalization Module - Visits to Health Care Providers - Acute and Continuation Phases
Description: Measures direct and indirect costs. Direct costs include inpatient and outpatient costs, while indirect costs include lost days of work and caregiver time spent with patients. Patients self-report on number of days over the past month that they have been either late to work, missed work, or missed usual activities due to symptoms.
Time Frame: Week 0 through Week10 (Acute) through Week 34 (Continuation)
Population: Number of enrolled patients in Acute Phase and number who entered Continuation Phase who indicated they had visits to specified health care provider. Intent to Treat analysis. Note: "Other Mental Health Care Worker" wasn't included in table (1 patient in Acute). "Other Health Care Worker" wasn't included in table (2 patients in Continuation).
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 514 | 413
visits
  Primary Health Care Provider Visits (N=94,N=99) | -0.00 (0.03) | -0.00 (0.03)
  Psychiatrist Visits (N=91,N=65) | 0.03 (0.03) | -0.03 (0.04)
  Psychologist/Therapist Visits (N=19,N=11) | 0.01 (0.04) | -0.00 (0.06)
  Other Specialist Physician Visits (N=42,N=38) | -0.00 (0.02) | 0.01 (0.03)
  Other (Specified by Patient) Visits (N=3,N=3) | 0.04 (0.07) | -0.07 (0.10)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.838, t-test, 2 sided — P-value for change in number of Primary Health Care Provider Visits in Acute Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for change in number of Psychiatrist visits in Acute Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 3: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.236, t-test, 2 sided — P-value for change in number of Psychologist/Therapist visits in Acute Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 4: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.145, t-test, 2 sided — P-value for change in number of Other Specialist Physician visits in Acute Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 5: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.423, t-test, 2 sided — P-value for change in number of Other (Specified by Patient) visits in Acute Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 6: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.325, t-test, 2 sided — P-value for change in number of Primary Health Care Provider visits in Continuation Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 7: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for change in number of Psychiatrist visits in Continuation Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 8: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.915, t-test, 2 sided — P-value for change in number of Psychologist/Therapist visits in Continuation Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 9: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.223, t-test, 2 sided — P-value for change in number of Other Specialist Physician visits in Continuation Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 10: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.362, t-test, 2 sided — P-value for change in number of Other (Specified by Patient) visits in Continuation Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

22. Secondary Outcome: Resource Utilization and Hospitalization Module - Visits to Health Care Providers - Maintenance Phase
Description: as for outcome 21
Time Frame: Week 34 through Week 86 (Maintenance Phase)
Population: Number of randomized patients who indicated they had visits to specified health care provider. Intent to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: visits
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 146 | 142
visits
  Primary Health Care Provider Visits (N=47,N=47) | -0.00 (0.00) | -0.00 (0.00)
  Psychiatrist Visits (N=33,N=23) | -0.01 (0.00) | -0.01 (0.01)
  Psychologist/Therapist Visits (N=8,N=7) | -0.02 (0.01) | -0.01 (0.01)
  Other Specialist Physician Visits (N=25,N=25) | 0.00 (0.01) | -0.00 (0.00)
  Other (Specified by Patient) Visits (N=5,N=3) | 0.04 (0.02) | 0.00 (0.00)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.462, t-test, 2 sided — P-value for pairwise comparison of means for change from baseline to endpoint in Primary Health Care Provider visits
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.668, t-test, 2 sided — P-value for pairwise comparison of means for change from baseline to endpoint in Psychiatrist visits
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.746, t-test, 2 sided — P-value for pairwise comparison of means for change from baseline to endpoint in Psychologist/Therapist visits
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.511, t-test, 2 sided — P-value for pairwise comparison of means for change from baseline to endpoint in Other Specialist Physician visits
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.271, t-test, 2 sided — P-value for pairwise comparison of means for change from baseline to endpoint in Other (Specified by Patient) Provider visits

23. Secondary Outcome: Resource Utilization and Hospitalization Module - Change From Baseline to Endpoint in Average Number of Hours Worked in a Week - Acute and Continuation Phases
Description: as for outcome 21
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: Number of enrolled patients in the Acute Phase who work for pay. Number of patients who entered the Continuation Phase who work for pay. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 224 | 196
hours
  Average Number of Hours Worked In a Week Baseline | 0.36 (0.10) | 0.36 (0.10)
  Change in Average Number of Hours Worked In a Week | 0.00 (0.06) | 0.01 (0.08)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.506, t-test, 2 sided — P-value for Change in Average Number of Hours Worked In a Week in Acute Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.057, t-test, 2 sided — P-value for Change in Average Number of Hours Worked In a Week in Continuation Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

24. Secondary Outcome: Resource Utilization and Hospitalization Module - Change From Baseline to Endpoint in Average Number of Hours Worked in a Week - Maintenance Phase
Description: as for outcome 21
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: Number of randomized patients who work for pay. Intent to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 87 | 83
hours | -0.00 (0.01) | -0.00 (0.01)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.826, t-test, 2 sided

25. Secondary Outcome: Resource Utilization and Hospitalization Module - Change From Baseline to Endpoint in Number of Missed Paid Work Hours - Acute and Continuation Phase
Description: as for outcome 21
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: Number of enrolled patients in the Acute Phase who work for pay and missed work due to illness. Number of patients who entered the Continuation Phase who work for pay and missed work due to illness. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Duloxetine - Acute; Duloxetine - Continuation Phase: duloxetine 60-120 mg QD
Arm/Group | Duloxetine - Acute | Duloxetine - Continuation Phase
Number analyzed (Participants) | 64 | 29
hours
  Number of Missed Paid Work Hours Baseline | 1.77 (2.07) | 2.67 (2.27)
  Change in Number of Missed Paid Work Hours | 0.46 (2.25) | -0.52 (2.01)
Statistical Analysis 1: Comparison: Duloxetine - Acute; Test type: Superiority or Other; p = 0.105, t-test, 2 sided — P-value for Change in Number of Missed Paid Work Hours in Acute Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.174, t-test, 2 sided — P-value for Change in Number of Missed Paid Work Hours in Continuation Phase; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

26. Secondary Outcome: Resource Utilization and Hospitalization Module - Change From Baseline to Endpoint in Number of Missed Paid Work Hours - Maintenance Phase
Description: as for outcome 21
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: Number of randomized patients who work for pay and missed work due to illness. Intent to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 13 | 16
hours | 0.27 (0.28) | -0.75 (0.35)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.037, t-test, 2 sided

27. Secondary Outcome: Change From Baseline to Endpoint in Arizona Sexual Experience Scale (ASEX) - Acute and Continuation Phases (Males)
Description: A 5-item patient-rated scale measuring 5 domains: sexual drive, arousal (subjective excitement), lubrication/erection (physiological excitement), ability to reach orgasm, orgasm satisfaction. Higher score means worse dysfunction. Total score range is 5-30.
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: Number of male enrolled patients in the Acute Phase with a baseline and at least one non-missing post-baseline measurement. Number of male patients who entered Continuation Phase with a baseline and have at least 1 post-baseline measurement. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 136 | 109
units on a scale
  Sum Items 1 to 5 Baseline (N=117,N=97) | 17.57 (4.88) | 17.26 (4.51)
  Sum Items 1 to 5 Change to Endpoint | 0.13 (5.08) | -0.67 (3.97)
  Sum Items 1&2 Baseline (N=135, N=109) | 7.47 (2.19) | 7.16 (1.96)
  Sum Items 1&2 Change to Endpoint | -0.19 (2.32) | -0.39 (1.76)
  Item 1-Sex Drive Baseline (N=136,N=109) | 3.91 (1.20) | 3.68 (1.14)
  Item 1-Sex Drive Change to Endpoint | -0.15 (1.30) | -0.21 (1.10)
  Item 2-Arousal Baseline (N=135, N=109) | 3.56 (1.11) | 3.48 (0.95)
  Item 2-Arousal Change to Endpoint | -0.02 (1.17) | -0.18 (0.83)
  Item 3-Lubrication/Erection Baseline (N=124,N=99) | 3.43 (1.13) | 3.27 (1.02)
  Item 3-Lubrication Change to Endpoint | -0.02 (1.15) | -0.04 (0.94)
  Item 4-Orgasm Baseline (N=120,N=98) | 3.38 (1.10) | 3.60 (1.03)
  Item 4-Orgasm Change to Endpoint | 0.32 (1.30) | -0.15 (1.01)
  Item 5-Satisfaction Baseline (N=118,N=97) | 3.36 (1.17) | 3.32 (1.20)
  Item 5-Satisfaction Change to Endpoint | 0.05 (1.29) | -0.15 (1.05)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.785, t-test, 2 sided — P-value for Sum Items 1 to 5 Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.354, t-test, 2 sided — P-value for Sum Items 1&2 Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 3: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.170, t-test, 2 sided — P-value for Item 1-Sex Drive Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 4: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.825, t-test, 2 sided — P-value for Item 2-Arousal Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 5: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.877, t-test, 2 sided — P-value for Item 3-Vaginal Lubrication/Penile Erection Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 6: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.009, t-test, 2 sided — P-value for Item 4-Orgasm Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 7: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.670, t-test, 2 sided — P-value for Item 5-Satisfaction Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 8: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.100, t-test, 2 sided — P-value for Sum Items 1 to 5 Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 9: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.021, t-test, 2 sided — P-value for Sum Items 1&2 Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 10: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.047, t-test, 2 sided — P-value for Item 1-Sex Drive Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 11: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.023, t-test, 2 sided — P-value for Item 2-Arousal Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 12: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.668, t-test, 2 sided — P-value for Item 3-Vaginal Lubrication/Penile Erection Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 13: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.136, t-test, 2 sided — P-value for Item 4-Orgasm Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 14: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.152, t-test, 2 sided — P-value for Item 5-Satisfaction Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

28. Secondary Outcome: Change From Baseline to Endpoint in Arizona Sexual Experience Scale (ASEX) - Acute and Continuation Phases (Females)
Description: as for outcome 27
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: Number of female enrolled patients in the Acute Phase with a baseline and at least one non-missing post-baseline measurement. Number of female patients who entered Continuation Phase with a baseline and have at least 1 post-baseline measurement. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 286 | 239
units on a scale
  Sum Items 1 to 5 Baseline (N=220,N=197) | 21.41 (5.17) | 19.31 (4.94)
  Sum Items 1 to 5 Change to Endpoint | -1.31 (3.91) | -0.99 (4.38)
  Sum Items 1&2 Baseline (N=285,N=239) | 9.31 (2.08) | 8.42 (2.28)
  Sum Items 1&2 Change to Endpoint | -0.69 (1.91) | -0.56 (1.92)
  Item 1-Sex Drive Baseline (N=286,N=239) | 4.92 (1.12) | 4.34 (1.20)
  Item 1-Sex Drive Change to Endpoint | -0.46 (1.05) | -0.31 (1.09)
  Item 2-Arousal Baseline (N=286,N=239) | 4.40 (1.13) | 4.08 (1.19)
  Item 2-Arousal Change to Endpoint | -0.22 (1.07) | -0.25 (1.02)
  Item 3-Lubrication/Erection Baseline (N=224,N=198) | 3.97 (1.26) | 3.57 (1.20)
  Item 3-Lubrication/Erection Change to Endpoint | -0.19 (0.98) | -0.10 (1.07)
  Item 4-Orgasm Baseline (N=224,N=198) | 4.33 (1.19) | 4.06 (1.08)
  Item4-Orgasm Change to Endpoint | -0.13 (1.02) | -0.28 (1.05)
  Item 5-Satisfaction Baseline (N=226,N=198) | 3.93 (1.39) | 3.58 (1.31)
  Item 5-Satisfaction Change to Endpoint | -0.18 (1.18) | -0.10 (1.32)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Sum Items 1 to 5 Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Sum Items 1&2 Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 3: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Item 1-Sex Drive Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 4: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Item 2-Arousal Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 5: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.005, t-test, 2 sided — P-value for Item 3-Vaginal Lubrication/Penile Erection Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 6: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.050, t-test, 2 sided — P-value for Item 4-Orgasm Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 7: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.022, t-test, 2 sided — P-value for Item 5-Satisfaction Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 8: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.002, t-test, 2 sided — P-value for Sum Items 1 to 5 Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 9: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Sum Items 1&2 Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 10: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Item 1-Sex Drive Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 11: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Item 2-Arousal Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 12: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.186, t-test, 2 sided — P-value for Item 3-Vaginal Lubrication/Penile Erection Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 13: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Item 4-Orgasm Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 14: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.308, t-test, 2 sided — P-value for Item 5-Satisfaction Change to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

29. Secondary Outcome: Change From Baseline to Endpoint in Arizona Sexual Experience Scale (ASEX) - Maintenance Phase (Males)
Description: as for outcome 27
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: N=Number of male randomized patients with non-missing baseline and at least one non-missing post-baseline measurement. Male patients who have been sexually active in the previous month respond to Items 3-5. Intent to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 39 | 29
units on a scale
  Change from Baseline: Sum Items 1 to 5 (N=35,N=29) | -0.97 (0.47) | -0.77 (0.58)
  Change from Baseline: Sum Items 1&2 (N=39,N=29) | -0.25 (0.22) | 0.03 (0.28)
  Item 1-Sex Drive (N=39,N=29) | -0.17 (0.13) | -0.02 (0.17)
  Item 2-Arousal (N=39,N=29) | -0.09 (0.12) | 0.07 (0.15)
  Item 3-Lubrication/Erection (N=38,N=29) | -0.32 (0.14) | -0.10 (0.17)
  Item 4-Orgasm (N=36,N=29) | -0.08 (0.14) | -0.43 (0.17)
  Item 5-Satisfaction (N=35,N=29) | -0.13 (0.11) | -0.04 (0.13)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.773, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for the Sum of Items 1 to 5
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.405, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for the Sum of Items 1 and 2
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.443, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for Item 1-Sex Drive
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.384, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for Item 2-Arousal
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.268, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for Item 3-Vaginal Lubrication/Penile Erection
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.093, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for Item 4-Orgasm
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.566, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for Item 5-Satisfaction

30. Secondary Outcome: Change From Baseline to Endpoint in Arizona Sexual Experience Scale (ASEX) - Maintenance Phase (Females)
Description: as for outcome 27
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: N=Number of female randomized patients with non-missing baseline and at least one non-missing post-baseline measurement. Female patients who have been sexually active in the previous month respond to Items 3-5. Intent to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 77 | 79
units on a scale
  Change from Baseline:Sum Items 1 to 5 (N=63,N=66) | -0.65 (4.14) | -0.47 (4.34)
  Change from Baseline:Sum Items 1&2 (N=77,N=79) | -0.19 (1.90) | 0.34 (1.91)
  Item 1 - Sex Drive (N=77,N=79) | -0.08 (1.11) | 0.18 (1.07)
  Item 2 - Arousal (N=77,N=79) | -0.12 (0.95) | 0.16 (1.06)
  Item 3 - Lubrication/Erection (N=63,N=67) | -0.21 (0.92) | -0.15 (1.21)
  Item 4 - Orgasm (N=63,N=67) | -0.10 (0.96) | -0.15 (1.06)
  Item 5 - Satisfaction (N=63,N=67) | -0.05 (1.25) | -0.40 (1.21)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.979, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for the Sum of Items 1 to 5
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.132, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for the Sum of Items 1 and 2
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.180, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for Item 1-Sex Drive
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.163, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for Item 2-Arousal
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.844, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for Item 3-Vaginal Lubrication/Penile Erection
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.609, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for Item 4-Orgasm
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.071, t-test, 2 sided — P-value for pairwise comparison Least Squares Mean change from baseline for Item 5-Satisfaction

31. Secondary Outcome: Vital Signs - Change From Baseline to Endpoint in Weight - Acute and Continuation Phases
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 503 | 412
kilograms
  Weight Baseline | 74.74 (16.25) | 74.22 (15.89)
  Weight Change from Baseline to Endpoint | -0.69 (2.12) | 0.88 (3.29)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Weight Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Weight Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

32. Secondary Outcome: Vital Signs - Change From Baseline to Endpoint in Weight - Maintenance Phase
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: Number of randomized patients with baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 145 | 142
kilograms | 0.88 (0.36) | 0.39 (0.37)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.314, t-test, 2 sided

33. Secondary Outcome: Vital Signs - Change From Baseline to Endpoint in Pulse - Acute and Continuation Phases
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 502 | 412
beats per minute
  Pulse Baseline | 71.76 (9.26) | 72.79 (9.50)
  Pulse Change from Baseline to Endpoint | 1.42 (9.18) | 1.75 (10.39)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Pulse Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value for Pulse Change from Baseline to Endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

34. Secondary Outcome: Vital Signs - Change From Baseline to Endpoint in Pulse - Maintenance Phase
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: Number of randomized patients with baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 145 | 142
beats per minute | -1.86 (0.76) | -1.72 (0.78)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.891, t-test, 2 sided

35. Secondary Outcome: Vital Signs - Change From Baseline to Endpoint in Blood Pressure - Acute and Continuation Phases
Time Frame: Week 0 and Week 10 (Acute) and Week 34 (Continuation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Duloxetine - Acute Phase | Duloxetine - Continuation Phase
Number analyzed (Participants) | 503 | 412
mm Hg
  Systolic Blood Pressure Baseline | 125.03 (14.65) | 124.72 (13.84)
  Systolic Blood Pressure Change to Endpoint | 0.25 (12.62) | 0.77 (12.83)
  Diastolic Blood Pressure Baseline | 77.52 (9.54) | 78.28 (9.19)
  Diastolic Blood Pressure Change to Endpoint | 0.72 (8.68) | -0.57 (9.18)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.659, t-test, 2 sided — P-value for systolic blood pressure change to endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 2: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = 0.064, t-test, 2 sided — P-value for diastolic blood pressure change to endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 3: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.224, t-test, 2 sided — P-value for systolic blood pressure change to endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero
Statistical Analysis 4: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = 0.210, t-test, 2 sided — P-value for diastolic blood pressure change to endpoint; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

36. Secondary Outcome: Vital Signs - Change From Baseline to Endpoint in Blood Pressure - Maintenance Phase
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: Number of randomized patients with baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 145 | 142
mm Hg
  Change from Baseline: Systolic Blood Pressure | 1.70 (13.44) | -1.11 (11.59)
  Change from Baseline: Diastolic Blood Pressure | -0.23 (9.72) | -0.11 (8.69)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.134, t-test, 2 sided — P-value for Change from Baseline: systolic blood pressure
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.816, t-test, 2 sided — P-value for Change from Baseline: diastolic blood pressure

37. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Albumin - Acute Phase
Time Frame: Week 0 and Week 10
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: grams per Liter
Arm/Group | Duloxetine - Acute Phase
Number analyzed (Participants) | 430
grams per Liter
  Baseline | 43.05 (3.31)
  Change to Endpoint | -0.61 (2.90)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < .001, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

38. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Calcium - Acute Phase
Time Frame: Week 0 and Week 10
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: millimoles per Liter
Arm/Group | Duloxetine - Acute Phase
Number analyzed (Participants) | 435
millimoles per Liter
  Baseline | 2.46 (0.10)
  Change to Endpoint | -0.01 (0.10)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = .007, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

39. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Chloride - Acute Phase
Time Frame: Week 0 and Week 10
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: millimoles per Liter
Arm/Group | Duloxetine - Acute Phase
Number analyzed (Participants) | 435
millimoles per Liter
  Baseline | 103.73 (2.66)
  Change to Endpoint | -0.29 (2.81)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = .035, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

40. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Eosinophils - Acute Phase
Time Frame: Week 0 and Week 10
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: Giga per Liter
Arm/Group | Duloxetine - Acute Phase
Number analyzed (Participants) | 423
Giga per Liter
  Baseline | 0.13 (0.09)
  Change to Endpoint | 0.01 (0.09)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = .021, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

41. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Gamma-Glutamyl Transferase - Acute Phase
Time Frame: Week 0 and Week 10
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | Duloxetine - Acute Phase
Number analyzed (Participants) | 434
Units per Liter
  Baseline | 29.25 (36.30)
  Change to Endpoint | -5.12 (20.53)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < .001, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

42. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Hematocrit - Acute Phase
Time Frame: Week 0 and Week 10
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: actual count
Arm/Group | Duloxetine - Acute Phase
Number analyzed (Participants) | 416
actual count
  Baseline | 0.43 (0.04)
  Change to Endpoint | -0.00 (0.03)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = .019, t-test, 2 sided — The mean change to endpoint of -0.00 indicates that on average, endpoint score decreased from baseline score by less than 0.005 units; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

43. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Hemoglobin - Acute Phase
Time Frame: Week 0 and Week 10
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: millimoles per Liter
Arm/Group | Duloxetine - Acute Phase
Number analyzed (Participants) | 423
millimoles per Liter
  Baseline | 8.81 (0.80)
  Change to Endpoint | -0.07 (0.48)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = .005, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

44. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Platelet Count - Acute Phase
Time Frame: Week 0 and Week 10
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: Giga per Liter
Arm/Group | Duloxetine - Acute Phase
Number analyzed (Participants) | 422
Giga per Liter
  Baseline | 261.08 (60.89)
  Change to Endpoint | 4.23 (40.22)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p = .031, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

45. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Sodium - Acute Phase
Time Frame: Week 0 and Week 10
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: millimoles per Liter
Arm/Group | Duloxetine - Acute Phase
Number analyzed (Participants) | 435
millimoles per Liter
  Baseline | 141.21 (2.65)
  Change to Endpoint | -0.64 (2.96)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < .001, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

46. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Total Protein - Acute Phase
Time Frame: Week 0 and Week 10
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: grams per Liter
Arm/Group | Duloxetine - Acute Phase
Number analyzed (Participants) | 435
grams per Liter
  Baseline | 73.59 (4.40)
  Change to Endpoint | -1.18 (4.11)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < .001, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

47. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Uric Acid - Acute Phase
Time Frame: Week 0 and Week 10
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: micromoles per Liter
Arm/Group | Duloxetine - Acute Phase
Number analyzed (Participants) | 435
micromoles per Liter
  Baseline | 297.05 (81.68)
  Change to Endpoint | -10.64 (49.42)
Statistical Analysis 1: Comparison: Duloxetine - Acute Phase; Test type: Superiority or Other; p < .001, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

48. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Albumin - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: grams per Liter
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 390
grams per Liter
  Baseline | 42.43 (3.04)
  Change to Endpoint | -0.57 (2.81)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < .001, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

49. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Bicarbonate, HCO3 - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: millimoles per Liter
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 389
millimoles per Liter
  Baseline | 24.41 (2.64)
  Change to Endpoint | 1.04 (2.93)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < .001, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

50. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Bilirubin, Direct - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: micromoles per Liter
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 388
micromoles per Liter
  Baseline | 2.03 (1.04)
  Change to Endpoint | -0.12 (0.85)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = .004, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

51. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Bilirubin, Total - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: micromoles per Liter
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 390
micromoles per Liter
  Baseline | 8.68 (5.10)
  Change to Endpoint | -0.50 (3.84)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = .010, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

52. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Calcium - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: millimoles per Liter
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 391
millimoles per Liter
  Baseline | 2.45 (0.10)
  Change to Endpoint | -0.01 (0.10)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = .003, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

53. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Erythrocyte Count - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: Tera per Liter
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 386
Tera per Liter
  Baseline | 4.74 (0.45)
  Change to Endpoint | -0.06 (0.25)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < .001, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

54. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Gamma-Glutamyl Transferase - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 392
Units per Liter
  Baseline | 24.13 (24.96)
  Change to Endpoint | 2.11 (17.11)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = .015, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

55. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Hematocrit - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: Actual count
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 384
Actual count
  Baseline | 0.42 (0.04)
  Change to Endpoint | -0.00 (0.03)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = .021, t-test, 2 sided — [p-value comment as in outcome 42, analysis 1]; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

56. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Hemoglobin - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: millimoles per Liter
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 386
millimoles per Liter
  Baseline | 8.73 (0.80)
  Change to Endpoint | -0.14 (0.47)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < .001, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

57. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Leukocyte Count - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: Giga per Liter
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 386
Giga per Liter
  Baseline | 6.40 (1.69)
  Change to Endpoint | 0.17 (1.57)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = .032, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

58. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Low Density Lipoprotein (LDL) Cholesterol (Direct) - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: millimoles per Liter
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 340
millimoles per Liter
  Baseline | 3.61 (1.07)
  Change to Endpoint | -0.14 (0.73)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < .001, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

59. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Mean Cell Hemoglobin - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: millimoles per Liter
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 384
millimoles per Liter
  Baseline | 20.73 (0.87)
  Change to Endpoint | -0.18 (0.99)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p < .001, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

60. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Mean Cell Volume (MCV) - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 384
femtoliters
  Baseline | 89.33 (5.10)
  Change to Endpoint | 0.45 (4.00)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = .028, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

61. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Monocytes - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: Giga per Liter
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 386
Giga per Liter
  Baseline | 0.35 (0.12)
  Change to Endpoint | 0.02 (0.12)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = .008, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

62. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Total Protein - Continuation Phase
Time Frame: Week 10 (baseline) and Week 34 (endpoint) (Continuation Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: grams per Liter
Arm/Group | Duloxetine - Continuation Phase
Number analyzed (Participants) | 392
grams per Liter
  Baseline | 72.47 (3.93)
  Change to Endpoint | -0.38 (3.77)
Statistical Analysis 1: Comparison: Duloxetine - Continuation Phase; Test type: Superiority or Other; p = .046, t-test, 2 sided; t-test assesses if within treatment mean changes from baseline to endpoint are significantly different from zero

63. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Alanine Aminotransferase (ALT) - Maintenance Phase
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 143 | 133
Units per Liter
  Baseline | 21.81 (11.56) | 22.12 (11.11)
  Change to Endpoint | 2.52 (15.40) | -0.38 (12.53)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.035, ANOVA — P-value for Change to Endpoint; Type II Sums of Squares from an analysis of variance (ANOVA) on the Ranks: Model = Pooled Investigator and Therapy

64. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Calcium - Maintenance Phase
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: millimoles per Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 143 | 133
millimoles per Liter
  Baseline | 2.43 (0.10) | 2.43 (0.08)
  Change to Endpoint | -0.04 (0.10) | -0.01 (0.09)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.011, ANOVA — P-value for Change to Endpoint; Type II Sums of Squares from an analysis of variance (ANOVA) on the Ranks: Model = Pooled Investigator and Therapy

65. Secondary Outcome: Statistically Significant Laboratory Measurements - Change From Baseline to Endpoint in Glucose - Maintenance Phase
Time Frame: Week 34 (baseline) and Week 86 (endpoint) (Maintenance Phase)
Population: Number of patients with a baseline and at least one non-missing post-baseline value. Intent to Treat analysis.
Measure: Mean (Standard Deviation); unit: millimoles per Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 120 | 112
millimoles per Liter
  Fasting Glucose Baseline (N=120,N=112) | 5.40 (0.72) | 5.47 (1.09)
  Fasting Glucose Change to Endpoint | 0.07 (0.71) | 0.03 (1.01)
  Non-Fasting Glucose Baseline (N=41,N=39) | 5.68 (0.91) | 5.74 (2.34)
  Non-Fasting Glucose Change to Endpoint | -0.20 (1.18) | 0.62 (1.67)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.744, ANOVA — P-value for fasting glucose change from baseline to endpoint; Type II Sums of Squares from an analysis of variance (ANOVA) on the Ranks: Model = Pooled Investigator and Therapy
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.030, ANOVA — P-value for non-fasting glucose change from baseline to endpoint; Type II Sums of Squares from an analysis of variance (ANOVA) on the Ranks: Model = Pooled Investigator and Therapy

66. Secondary Outcome: Treatment-Emergent Adverse Events Occurring in at Least 5 Percent of Participants -- Open-Label Acute Therapy Phase
Time Frame: Every Visit from Week 0 up to Week 10 (Acute)
Population: Treatment-Emergent Adverse Events (TEAE) occurring in at least 5% of patients. Intent to Treat analysis.
Measure: Number; unit: participants
Arm/Group | Duloxetine - Acute Phase
Number analyzed (Participants) | 514
participants
  Patients with >= 1 Adverse Event | 349
  Nausea | 150
  Headache | 79
  Dry mouth | 76
  Hyperhidrosis | 76
  Fatigue | 60
  Constipation | 48
  Dizziness | 41
  Diarrhoea | 38
  Vomiting | 28
  Insomnia | 27
  Decreased appetite | 26

67. Secondary Outcome: Treatment-Emergent Adverse Events Occurring in at Least 5 Percent of the Participants -- Open-Label Continuation Phase
Time Frame: Every Visit from Week 10 up to Week 34 (Continuation)
Population: Treatment-Emergent Adverse Events (TEAE) occurring in at least 5% of patients. Intent to Treat analysis.
Measure: Number; unit: participants
Groups:
- Duloxetine 60 mg: duloxetine 60 mg every day (QD) from Week 10 (baseline) to Week 34 (Endpoint)
- Duloxetine 90 mg: duloxetine 90 mg every day (QD) from Week 10 (baseline) to Week 34 (Endpoint)
- Duloxetine 120 mg: duloxetine 120 mg every day (QD) from Week 10 (baseline) to Week 34 (Endpoint)
Arm/Group | Duloxetine 60 mg | Duloxetine 90 mg | Duloxetine 120 mg
Number analyzed (Participants) | 175 | 128 | 110
participants
  Patients with >= 1 Adverse Event | 102 | 83 | 59
  Headache | 21 | 12 | 6
  Nasopharyngitis | 7 | 10 | 9
  Hyperhidrosis | 8 | 12 | 5
  Back pain | 7 | 4 | 8
  Diarrhoea | 10 | 6 | 2

ADVERSE EVENTS:
Groups:
- Placebo: Placebo
- Duloxetine 60 mg: Duloxetine 60 mg
- Duloxetine 90 mg: Duloxetine 90 mg
- Duloxetine 120 mg: Duloxetine 120 mg
Arm/Group | Placebo | Duloxetine 60 mg | Duloxetine 90 mg | Duloxetine 120 mg
Serious Adverse Events (participants affected / at risk) | 5 | 5 | 3 | 4
Other Adverse Events (participants affected / at risk) | 105 | 51 | 36 | 26
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Duloxetine 60 mg | Duloxetine 90 mg | Duloxetine 120 mg
Myocardial ischaemia (Cardiac disorders) | 0/142 (0) | 0/64 (0) | 0/45 (0) | 1/37 (1)
Diverticular perforation (Gastrointestinal disorders) | 0/142 (0) | 1/64 (1) | 1/45 (1) | 0/37 (0)
Abscess (Infections and infestations) | 0/142 (0) | 0/64 (0) | 1/45 (1) | 0/37 (0)
Endocarditis staphylococcal (Infections and infestations) | 0/142 (0) | 1/64 (1) | 0/45 (0) | 0/37 (0)
Pneumonia chlamydial (Infections and infestations) | 0/142 (0) | 0/64 (0) | 1/45 (1) | 0/37 (0)
Pyelonephritis (Infections and infestations) | 0/142 (0) | 0/64 (0) | 1/45 (1) | 0/37 (0)
Skin bacterial infection (Infections and infestations) | 0/142 (0) | 1/64 (1) | 0/45 (0) | 0/37 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1/142 (1) | 0/64 (0) | 0/45 (0) | 0/37 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1/142 (1) | 0/64 (0) | 0/45 (0) | 1/37 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/142 (1) | 1/64 (1) | 0/45 (0) | 0/37 (0)
Migraine (Nervous system disorders) | 0/142 (0) | 1/64 (1) | 0/45 (0) | 0/37 (0)
Transient ischaemic attack (Nervous system disorders) | 0/142 (0) | 0/64 (0) | 0/45 (0) | 1/37 (1)
Depression (Psychiatric disorders) | 0/142 (0) | 0/64 (0) | 0/45 (0) | 1/37 (1)
Major depression (Psychiatric disorders) | 1/142 (1) | 0/64 (0) | 0/45 (0) | 0/37 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/142 (1) | 0/64 (0) | 0/45 (0) | 0/37 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Duloxetine 60 mg | Duloxetine 90 mg | Duloxetine 120 mg
Palpitations (Cardiac disorders) | 2/142 (2) | 1/64 (1) | 3/45 (3) | 0/37 (0)
Abdominal pain (Gastrointestinal disorders) | 3/142 (3) | 5/64 (7) | 0/45 (0) | 1/37 (1)
Abdominal pain upper (Gastrointestinal disorders) | 4/142 (4) | 4/64 (5) | 1/45 (1) | 2/37 (2)
Constipation (Gastrointestinal disorders) | 6/142 (6) | 3/64 (3) | 3/45 (3) | 2/37 (2)
Diarrhoea (Gastrointestinal disorders) | 10/142 (12) | 3/64 (3) | 5/45 (7) | 1/37 (1)
Dry mouth (Gastrointestinal disorders) | 9/142 (9) | 5/64 (5) | 11/45 (14) | 4/37 (4)
Dyspepsia (Gastrointestinal disorders) | 4/142 (5) | 2/64 (2) | 4/45 (4) | 2/37 (2)
Nausea (Gastrointestinal disorders) | 10/142 (12) | 7/64 (8) | 5/45 (6) | 1/37 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 1/142 (1) | 0/64 (0) | 0/45 (0) | 2/37 (2)
Fatigue (General disorders) | 8/142 (8) | 4/64 (4) | 7/45 (9) | 4/37 (4)
Pain (General disorders) | 2/142 (2) | 0/64 (0) | 3/45 (3) | 0/37 (0)
Hypersensitivity (Immune system disorders) | 0/142 (0) | 1/64 (1) | 3/45 (4) | 0/37 (0)
Seasonal allergy (Immune system disorders) | 1/142 (1) | 0/64 (0) | 0/45 (0) | 2/37 (2)
Bronchitis (Infections and infestations) | 6/142 (8) | 2/64 (2) | 3/45 (3) | 1/37 (1)
Influenza (Infections and infestations) | 15/142 (15) | 4/64 (4) | 2/45 (4) | 1/37 (1)
Nasopharyngitis (Infections and infestations) | 18/142 (26) | 10/64 (16) | 6/45 (8) | 3/37 (3)
Blood creatine phosphokinase increased (Investigations) | 4/142 (4) | 0/64 (0) | 0/45 (0) | 2/37 (2)
Electrocardiogram T wave abnormal (Investigations) | 0/142 (0) | 0/64 (0) | 1/45 (1) | 3/37 (3)
Weight increased (Investigations) | 3/142 (3) | 2/64 (2) | 4/45 (4) | 1/37 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5/142 (7) | 1/64 (2) | 3/45 (7) | 3/37 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 14/142 (14) | 8/64 (8) | 9/45 (10) | 5/37 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 1/142 (1) | 0/64 (0) | 2/45 (2) | 2/37 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1/142 (1) | 2/64 (2) | 1/45 (1) | 2/37 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6/142 (7) | 2/64 (2) | 2/45 (2) | 2/37 (5)
Dizziness (Nervous system disorders) | 12/142 (13) | 4/64 (4) | 2/45 (2) | 1/37 (1)
Headache (Nervous system disorders) | 30/142 (35) | 21/64 (28) | 11/45 (14) | 3/37 (4)
Migraine (Nervous system disorders) | 5/142 (6) | 2/64 (9) | 1/45 (1) | 2/37 (2)
Paraesthesia (Nervous system disorders) | 3/142 (3) | 1/64 (1) | 5/45 (7) | 1/37 (1)
Anxiety (Psychiatric disorders) | 7/142 (11) | 1/64 (1) | 1/45 (2) | 3/37 (3)
Insomnia (Psychiatric disorders) | 20/142 (22) | 4/64 (4) | 3/45 (3) | 2/37 (2)
Pollakiuria (Renal and urinary disorders) | 4/142 (4) | 0/64 (0) | 0/45 (0) | 2/37 (2)
Ejaculation delayed (Reproductive system and breast disorders) | 3/142 (3) | 1/64 (1) | 0/45 (0) | 2/37 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2/142 (2) | 0/64 (0) | 1/45 (1) | 2/37 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5/142 (7) | 4/64 (5) | 0/45 (0) | 0/37 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 19/142 (19) | 5/64 (5) | 13/45 (13) | 5/37 (6)
Hypertension (Vascular disorders) | 6/142 (6) | 1/64 (1) | 4/45 (4) | 1/37 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days